CLINICAL TRIAL: NCT02035059
Title: Predictability of Gestational Diabetes Mellitus in First and Second Trimester, Using Novel Biomarkers, and the Development of New Biomarkers by Quantitative Proteomic Analysis
Brief Title: Predictability of Gestational Diabetes Mellitus in First and Second Trimester
Acronym: GDMPredict
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University Hospital, Zürich (Other); Cantonal Hospital of Aarau, Switzerland (Other); Vienna General Hospital (Other); Paracelsus Medical University (Other); University Hospital Freiburg (Other)
Responsible Party: Sponsor
Other Study IDs: EKBB195/13
Record Dates: First submitted 2014-01-12; First posted 2014-01-14 (Estimated); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Pregnancy; Gestational Diabetes Mellitus
Keywords: Oral Glucose Tolerance Test; Fibronectin; Adiponectin; Copeptin; Cortisol
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Insipidus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood Saliva
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Women with/without gestational diabetes: Women with/without gestational diabetes diagnosed by clinically routine 75 g oral glucose tolerance testing

SUMMARY:
The objective of the study is, if an early oral glucose tolerance test combined with maternal history, condition and multiple biomarker analysis can be used to detect gestational diabetes mellitus in the first trimester (12-14 weeks of gestation).

DETAILED DESCRIPTION:
It is the investigators' aim to prospectively examine an extended form of the current 1st trimester screening test for the detection of foetal aneuploidy, in order to ascertain whether this can also be used for the detection of patients at-risk for gestational diabetes mellitus. For this purpose the investigators will include a combination of new markers in a multiplex bio-array manner in conjunction with an early oral glucose tolerance test. A nested case-control proteomic analysis will be performed in a retrospective manner at the completion of this study in order to develop more specific biomarker panels.

The primary outcome will be development of gestational diabetes mellitus in the second or third trimester.

The secondary endpoints are the delivery outcome, neonatal morbidity, neonatal mortality, maternal morbidity and costs.

ELIGIBILITY:
Inclusion Criteria:

* Healthy singleton pregnancies
* Women at least 18 years old and not under guardianship

Exclusion Criteria:

* Maternal diseases like hypertension, diabetes mellitus and chronic disease, known infection like hepatitis or human immunodeficiency virus
* Maternal history of hypertensive diseases in previous pregnancy and now under prophylactic acetylsalicylate treatment
* Foetal genetic, chromosomal or intervention-requiring morphologic abnormalities

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant Women
Sampling Method: Non-Probability Sample
Enrollment: 820 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Development of Gestational Diabetes in second/third trimester | 24-28 weeks of gestation
  Development of gestational diabetes in 24-28 weeks of gestation by pathological values in oral glucose tolerance test 75g

CONTACTS AND LOCATIONS:
Overall Officials: Evelyn Huhn, MD, Study Director — Women's Hospital, University Basel; Irene Hösli, MD, Principal Investigator — Women's Hospital, University Basel
Locations (1):
- Women's Hospital, University Basel, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Derived] Huhn EA, Kotzaeridi G, Fischer T, Todesco Bernasconi M, Richter AS, Kunze M, Dolzlmuller E, Jaksch-Bogensperger H, Weidinger L, Eppel D, Ochsenbein-Koelble N, Baz E, Winzeler B, Tura A, Stach H, Schafer G, van Breda SV, Vokalova L, Hoesli I, Gobl CS. The utility of early gestational OGTT and biomarkers for the development of gestational diabetes mellitus: an international prospective multicentre cohort study. Diabetologia. 2025 Nov;68(11):2511-2522. doi: 10.1007/s00125-025-06517-0. Epub 2025 Aug 16. PMID 40817933
- [Derived] Huhn EA, Gobl CS, Fischer T, Todesco Bernasconi M, Kreft M, Kunze M, Vogt DR, Dolzlmuller E, Jaksch-Bogensperger H, Heldstab S, Eppel W, Husslein P, Ochsenbein Kolble N, Richter A, Baz E, Winzeler B, Hoesli I. Sensitivity, specificity, and diagnostic accuracy of WHO 2013 criteria for diagnosis of gestational diabetes mellitus in low risk early pregnancies: international, prospective, multicentre cohort study. BMJ Med. 2023 Sep 13;2(1):e000330. doi: 10.1136/bmjmed-2022-000330. eCollection 2023. PMID 37720695
- [Derived] Huhn EA, Fischer T, Gobl CS, Todesco Bernasconi M, Kreft M, Kunze M, Schoetzau A, Dolzlmuller E, Eppel W, Husslein P, Ochsenbein-Koelble N, Zimmermann R, Baz E, Prompeler H, Bruder E, Hahn S, Hoesli I. Screening of gestational diabetes mellitus in early pregnancy by oral glucose tolerance test and glycosylated fibronectin: study protocol for an international, prospective, multicentre cohort trial. BMJ Open. 2016 Oct 12;6(10):e012115. doi: 10.1136/bmjopen-2016-012115. PMID 27733413